CLINICAL TRIAL: NCT02420158
Title: Sympatho-vagal Balance in Patients With Irritable Bowel Syndrome, and Evaluation of a Transcutaneous Vagal Nerve Electrical Stimulation on Symptoms and Quality of Life
Brief Title: Trans-cutaneous Vagal Nerve Electrical Stimulation and Irritable Bowel Syndrome
Acronym: StVSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.844
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2019-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Vagal nerve stimulation; Quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vagal nerve stimulation (Experimental): Trans-cutaneous vagal nerve electrical stimulation during 6 months
  Interventions: Device: Trans-cutaneous vagal nerve electrical stimulation

INTERVENTIONS:
Device: Trans-cutaneous vagal nerve electrical stimulation

SUMMARY:
This pilot study plan to investigate the sympathovagal balance in women affected by Irritable Bowel Syndrome (IBS), and to evaluate the effect of 6 months of trans-cutaneous vagal nerve electrical stimulation on digestive physiology (intestinal transit time, intestinal mucosal permeability, systemic and local inflammation), symptoms and quality of life.

The safety of the electrical stimulation of the left vagal nerve will also be evaluated.

Ten women, age between 18 and 60, will be included.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-60,
* clinical Rome III criteria for IBS

Exclusion Criteria:

* pregnancy,
* low intensity symptoms (Francis score between 75-150)
* IBD, coeliac disease
* past history of abdominal surgery (appendectomy and cholecystectomy allowed)
* chronic use of analgesics, anti-depressants

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Improvement of clinical symptoms of IBS, based on the evolution of symptom score (Francis) and symptom scale (UCLA-SSS) | 3 and 6 months after the beginning of electrical stimulation

SECONDARY OUTCOMES:
Safety and tolerance of trans-cutaneous nerve stimulation as measured by any symptom occurring in relation with electrical stimulation, number of hours per day of system use | 6 months
  Any symptom occurring in relation with electrical stimulation, number of hours per day of system use
Evolution of digestive physiology during vagal nerve stimulation | 3 and 6 months
  Digestive physiology is evaluated by intestinal transit time with Smartpill capsule, lactuose/mannitol intestinal permeability test, fecal calprotectin and blood cytokines
Effect of vagal nerve stimulation on quality of life | 3 and 6 months
  Quality of life and psychological questionnaires
Evaluation of sympatho-vagal balance | 0, 3 and 6 months
  Measurement by nocturnal EKG Holter of the variability of the interval RR, as a marker of the sympatho-vagal balance

CONTACTS AND LOCATIONS:
Overall Officials: François MION, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Clinique Universitaire d'Hépato-Gastroentérologie - CHU de Grenoble, Grenoble
  - Service d'Exploration Fonctionnelle Digestive - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon

REFERENCES:
- [Result] Short Communication BIOELECTRONICS IN MEDICINE Volume 3, 2020 - Issue 1 - Pages 5-12 Transcutaneous auricular vagus nerve stimulation for the treatment of irritable bowel syndrome: a pilot, open-label study Francois Mion*,1,2,3 , Sonia Pellissier4, Aur´ elien Garros1, Henri Damon1, Sabine Roman1,2,3 & Bruno Bonaz5,6,7 1Department of Digestive Physiology, Hospices Civils de Lyon, Lyon, France 2Department of Physiology, Universite´ de Lyon, Lyon, France 3Inserm U1032, LabTau, Lyon, France 4Universite´ Savoie Mont Blanc, Universite´ Grenoble Alpes, LIP/PC2S, 73000, Chambe´ ry 5Division of Hepato-Gastroenterology, CHU Grenoble Alpes, 38000 Grenoble, France 6Hepatogastroenterology, Universite´ Grenoble Alpes, Grenoble 7INSERM U1216, Grenoble Institute Neurosciences, Grenoble *Author for correspondence: francois.mion@chu-lyon.fr